CLINICAL TRIAL: NCT03187938
Title: Alkaline Phosphatase Level in Pregnancy and Its Association With Birth Weight
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-095
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Birth Weight Infants
Keywords: Alkaline Phosphatase; Pregnancy; Suboptimal fetal growth; Placental insufficiency; Low birth weight; IUGR
MeSH Terms: conditions — Placental Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women at 24-28 weeks gestation: Pregnant women, aged 18 and older, who are seen for their prenatal care and who are between 24w0d and 28w6d weeks gestation.Their alkaline phosphatase levels will be tested in this study.
  Interventions: Diagnostic Test: Testing of Alkaline Phosphatase Levels

INTERVENTIONS:
Diagnostic Test: Testing of Alkaline Phosphatase Levels — Testing of alkaline phosphatase levels at the time of the 24w0d to 28w6d week labs.

SUMMARY:
Alkaline phosphatase is known to be produced by syncytiotrophoblasts in the placenta and its levels are normally increased in pregnancy. Therefore, it would be reasonable to hypothesize that alkaline phosphatase would be low to low normal in cases of low birth weight / intrauterine growth restriction (IUGR)/ placental insufficiency.

DETAILED DESCRIPTION:
The purpose of this study will be to determine if alkaline phosphatase can be used as a predictor for suboptimal fetal growth, placental insufficiency and low birth weight (birth weight less than 2500 grams). It will also help determine if alkaline phosphatase can be used as a screening tool for low birth weight/IUGR at the time of the 24 to 28 week labs.

ELIGIBILITY:
Inclusion Criteria:

• Patients enrolled between 24w0d and 28w6d weeks gestational age will be included. The blood specimen of the patients enrolled will be held until delivery.

Exclusion Criteria:

* Multiple gestations
* Known congenital malformations (any, except Pyelectasis)
* Chronic hypertension
* Inflammatory bowel disease (IBD)
* Gall bladder disease
* Active bone disease (ie, skeletal dysplasia, healing fracture)
* Active liver disease (ie, hepatitis, cholestasis, cholelithiasis (gallstones))
* Pre-existing type 1 and 2 Diabetes
* Early-onset IUGR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women, aged 18 and older, who are seen for their prenatal care and who are between 24w0d and 28w6d weeks gestation.
Study Population: Pregnant women, aged 18 and older, who are seen for their prenatal care and who are between 24w0d and 28w6d weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Birth Weight at Delivery | At Delivery
  Birth Weight at Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Donna Lambers, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan TriHealth Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No